CLINICAL TRIAL: NCT03510156
Title: Treatment of Disruptive Behaviors in Fragile X Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The John Merck Fund (Unknown)
Responsible Party: Principal Investigator, Scott Hall, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36394
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Fragile X Syndrome; Disruptive Behavior
MeSH Terms: conditions — Fragile X Syndrome; Problem Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Behavioral: Behavior analytic treatment
- Observation (No Intervention)

INTERVENTIONS:
Behavioral: Behavior analytic treatment — Function-based treatment
  Arms: Treatment

SUMMARY:
Disruptive behaviors such as self-injury, aggression, and property destruction pose significant health-related issues to children diagnosed with fragile X syndrome (FXS), impacting the child's quality of life and causing significant distress to families.

Access to appropriate treatment for families is severely limited by factors such as cost of care, shortages of qualified treatment providers, and geographic spread of children with FXS across the country. To address these potential issues, the effectiveness of administering a standardized function-based behavioral treatment for problem behaviors in FXS will be evaluated using telemedicine. The proposed study intervention therefore offers a tremendous step forward in clinical research both in the field of FXS and in the field of developmental disabilities more broadly, and thus will have a significant impact on public health.

ELIGIBILITY:
Inclusion Criteria:

1. Child has a confirmed diagnosis of FXS (>200 CGG repeats on the FMR1 gene with evidence of aberrant methylation)
2. Child is male, between the ages of 3-10 years old
3. Child is reported to show self-injury, property destruction and/or aggression on at least a daily basis
4. The caregiver agrees to keep any therapies that the child receives (i.e., medications or other treatments) as stable as possible throughout involvement in the study
5. The family has a high-speed internet connection at home or lives in an area with 4G network coverage
6. Availability for one-hour daily telemedicine treatment sessions
7. Availability for in-home assessment totaling 8 hours across two consecutive days

Exclusion Criteria:

1. The child or caregiver has significant sensory impairments (e.g., blindness or deafness)
2. Non-English speaking
3. The child receives Applied Behavior Analysis services in excess of five hours per week
4. The child has a significant neurological condition (e.g., frequent seizures, brain injury, Tourette's syndrome) that would preclude participation
5. The child or caregiver has significant mobility issues
6. The child is currently participating in another research study that would preclude participation in the study

Ages: 3 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline level of problem behavior at 4, 8, 12 and 16 weeks | 0, 4, 8, 12, 16 weeks
  Aberrant Behavior Checklist - Community (ABC-C)

SECONDARY OUTCOMES:
Change from baseline level of treatment acceptability at 4, 8, 12 and 16 weeks | 0, 4, 8, 12, 16 weeks
  Treatment Acceptability Rating Form - Revised (TARF-R)

CONTACTS AND LOCATIONS:
Overall Officials: Scott S Hall, PhD, Principal Investigator — Stanford University
Locations (1):
- Department of Psychiatry and Behavioral Sciences, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall SS, Rodriguez AB, Jo B, Pollard JS. Long-term follow-up of telehealth-enabled behavioral treatment for challenging behaviors in boys with fragile X syndrome. J Neurodev Disord. 2022 Sep 30;14(1):53. doi: 10.1186/s11689-022-09463-9. PMID 36180840
- [Derived] Hall SS, Monlux KD, Rodriguez AB, Jo B, Pollard JS. Telehealth-enabled behavioral treatment for problem behaviors in boys with fragile X syndrome: a randomized controlled trial. J Neurodev Disord. 2020 Nov 20;12(1):31. doi: 10.1186/s11689-020-09331-4. PMID 33218305